CLINICAL TRIAL: NCT04946656
Title: A Study of SPG Block for Opioid Withdrawal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Diana Martinez, Professor of Psychiatry at Columbia University Irving Medical, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 7930
Record Dates: First submitted 2021-05-20; First posted 2021-07-01 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Sphenopalatine Ganglion Block

STUDY DESIGN:
Intervention Model Description: open label single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPG block (Experimental): The sphenopalatine ganglion will be blocked with bipuvacaine for this study
  Interventions: Procedure: sphenopalatine ganglion block

INTERVENTIONS:
Procedure: sphenopalatine ganglion block — The sphenopalatine ganglion will be blocked with bupivacaine for this study

SUMMARY:
Medication is the most efficacious treatment of an opioid use disorder, including methadone, buprenorphine, and naltrexone. However, many patients experience withdrawal symptoms, which prevents them from being successfully inducted onto medication for opioid use disorder. This study is a pilot study investigating whether blocking the SPG helps reduce withdrawal symptoms in OUD. This study does not involve treatment or induction onto medications. It is a proof of principal study only. We will recruit non-treatment seeking subjects with OUD who are admitted to the research unit for all procedures.

DETAILED DESCRIPTION:
The sphenopalatine ganglion (SPG) is a collection of neurons involved in autonomic regulation (which refers to bodily processes that are automatic like heart rate and blood pressure). Blocking the SPG is used to treat disorders, such as migraines or cluster headaches (short, severe headaches that occur together). The procedure will be performed by a doctor (specialized in ear, nose throat surgery) and would first involve the application of numbing nasal spray to both nostrils, which lasts about two hours and might reduce smell during that time. This is followed by an injection of a stronger numbing agent (similar to the type used by dentists) to the nerve bundles in the back of the nasal passages (one side at a time) via a tool, known as an endoscope which is a rigid tube with a camera on the end. The procedure is not painful. Previous studies have shown that clonidine, which inhibits the autonomic nervous system, is helpful for reducing the symptoms of opioid withdrawal. However, the dosing of clonidine is limited by side effects (lowered blood pressure and heart rate) and compliance. Furthermore, withdrawal is among the most significant barriers to substance treatment and ultimately overcoming a substance use disorder. Thus, we would like to explore whether a more targeted intervention would improve rates of successful acute detoxification while overcoming the aforementioned challenges of systemic side effects and compliance issues observed with the use of oral agents.

ELIGIBILITY:
Inclusion Criteria:

* Opioid Use Disorder, moderate to severe
* Ages 22 to 50
* Lives in New York City, able to travel for visits
* Willing to be admitted to an inpatient unit

Exclusion Criteria:

* Medical disorder, for who study participation could be deleterious (neurologic, cardiac, renal or infectious disease
* Hypertension: BP > 150/100
* Elevated liver function tests (AST, ALT) > 3x normal
* Having a painful medical illness for which opioids are needed (including upcoming surgery).

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
enrollment: percent screened subjects who enroll | 4 weeks
  We will measure the percent of screened participants who agree to enroll as part of the feasibility study
retention: percent enrolled subjects who complete | 4 weeks
  We will measure the percent of enrolled participants who complete the study as part of the feasibility study
tolerability: percent adverse events, if any | 4 weeks
  We will measure the percent of adverse events in this feasibility study, if any measured with the CTCAE grading system (rate 0 to 5)

CONTACTS AND LOCATIONS:
Locations (1):
- 1051 Riverside Drive, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No